CLINICAL TRIAL: NCT00502931
Title: A Systematic Review on the Accuracy and Reliability of a Hand-Held Indirect Calorimeter for Assessing Energy Needs in Adults & Children
Brief Title: A Systematic Review on the Accuracy and Reliability the BodyGem/MedGem Metabolic Devices
Status: Completed | Type: Observational
Sponsor: Microlife (Industry)
Other Study IDs: ML003
Record Dates: First submitted 2007-07-16; First posted 2007-07-18 (Estimated); Last update posted 2007-07-18 (Estimated); Status verified 2007-07

CONDITIONS: Resting Metabolic Rate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
With the number of individuals becoming overweight or obese, healthcare professionals are in need of accurate, reliable, and convenient tools to help personalize weight loss programs. Recently, a new indirect calorimeter (i.e. MedGem / BodyGem; aka "Gem") was introduced as a convenient solution to determine resting metabolic rate (RMR) for assessment of daily energy needs. Several validation and comparison studies were conducted to determine if the Gem device is accurate and reliable. The purpose of this study was to conduct a systematic review of previous studies that evaluated the accuracy and reliability of the Gem devices.

ELIGIBILITY:
Inclusion Criteria:

* Random or counterbalanced assignment of participants to eliminate measurement bias; similar subject positioning for both Gem and reference system measurement or adjustment to a measurement for positioning differences; and use of a measurement protocol that is similar to the established "best practice" guidelines for employing indirect calorimetry

Sex: All
Age Groups: Child, Adult, Older Adult
Dates: Start 2006-11

CONTACTS AND LOCATIONS:
Overall Officials: Scott O McDoniel, M.Ed., Principal Investigator — Microlife USA, Inc.
Locations (1):
- Microlife Health Solutions, Golden, Colorado, United States